CLINICAL TRIAL: NCT07031232
Title: Assessment of Peri-implant Soft Tissue Modifications Following the Use of Customized Healing Abutments on Subcrestally Placed Implants
Brief Title: Comparative Clinical Study of Conventional vs Customized Healing Abutments in Dental Implantology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Carlos Bernabeu Mira, Clinical Professor and Research Director in Oral Surgery and Implantology, Universitat de València, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-3494808
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Peri-implant Soft Tissue Healing; Soft Tissue Management in Subcrestal Dental Implants; Healing Abutment Influence on Gingival Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Healing Abutment Group (Experimental): Participants in this group will receive a conventional, prefabricated cylindrical titanium healing abutment placed immediately after implant surgery. The abutment will remain in place throughout the healing period, following a one abutment-one time protocol.
  Interventions: Procedure: Bone-Level Implant Placement with Transmucosal Abutment and One Abutment-One Time Protocol Using Healing Abutments
- Wide Healing Abutment Group (Experimental): Participants in this group will receive a prefabricated wide healing abutment with an increased diameter designed to provide broader mucosal support. The abutment will be placed immediately after surgery and will not be removed during healing.
  Interventions: Procedure: Bone-Level Implant Placement with Transmucosal Abutment and One Abutment-One Time Protocol Using Healing Abutments
- Customized Healing Abutment Group (Experimental): Participants in this group will receive a customized healing abutment fabricated with composite using a preform-phantoma. The abutment will replicate the desired emergence profile of the final prosthesis. It will be placed immediately after surgery and left in place during the healing phase.
  Interventions: Procedure: Bone-Level Implant Placement with Transmucosal Abutment and One Abutment-One Time Protocol Using Healing Abutments

INTERVENTIONS:
Procedure: Bone-Level Implant Placement with Transmucosal Abutment and One Abutment-One Time Protocol Using Healing Abutments — All participants will receive a single bone-level dental implant placed in a healed posterior site of the maxilla or mandible. The implants will be placed using a biological drilling protocol and inserted with a final torque of at least 30 Ncm. A 2 mm transmucosal one-piece abutment (mono-block) will be connected at the time of surgery, following a one abutment-one time philosophy.
  Each patient will receive a healing abutment immediately after implant placement according to their allocated study group (standard, wide, or customized). The assigned healing abutment will not be removed throughout the healing period. All procedures will be carried out under local anesthesia in a standard clinical setting.

SUMMARY:
This clinical study evaluates how different healing abutment designs influence the healing and preservation of the soft tissues surrounding dental implants. Healing abutments are temporary components placed on implants during the healing phase to help shape the gum tissue before placing the final crown or prosthesis. The way these components interact with the gum tissue may affect the long-term stability, volume, and aesthetics of the peri-implant soft tissue.

All participating patients will receive bone-level dental implants placed approximately 2 mm below the bone crest (subcrestal position). The study will include three groups of patients, each receiving a different type of healing abutment:

Group 1 (Control): will receive a standard cylindrical healing abutment.

Group 2: will receive a wide healing abutment with an enlarged base to support more soft tissue volume.

Group 3: will receive a customized healing abutment designed using digital intraoral scanning and CAD/CAM technology, intended to replicate the final prosthetic emergence profile.

The goal is to evaluate which type of healing abutment helps to preserve the natural volume and shape of the gum tissue most effectively during the healing period. The primary focus will be on measuring changes in soft tissue volume and thickness around the implants over time.

Participants will undergo digital intraoral scans before surgery and at 3, 6, and 12 months after implant placement. These scans will be used to assess how the gum tissue changes in response to each type of abutment using 3D analysis and software-based measurements.

This study is important because maintaining healthy and stable soft tissue around dental implants plays a crucial role in achieving successful, long-lasting, and aesthetically pleasing results. By understanding how healing abutment design affects tissue healing, clinicians may be better equipped to select the most appropriate healing protocol for each patient.

DETAILED DESCRIPTION:
Background and Rationale:

Peri-implant soft tissue health and stability are essential factors influencing the long-term success of dental implants, especially in terms of aesthetic outcomes and biological integration. A well-formed and stable mucosal seal around the implant protects the underlying bone, supports tissue homeostasis, and contributes to the overall functional and esthetic result of implant-supported prostheses.

Healing abutments are temporary components used during the transgingival healing phase to help shape the emergence profile and guide soft tissue adaptation prior to final prosthetic restoration. The design, diameter, and customization of the healing abutment may significantly affect peri-implant soft tissue volume, thickness, contour, and recession patterns. Recent research has suggested that minimizing disruption to the peri-implant mucosa (i.e., using a one abutment-one time approach) and optimizing soft tissue support during healing can result in improved tissue preservation and enhanced esthetic outcomes.

However, there is limited clinical evidence comparing the effect of different healing abutment designs-particularly standard, wide, and customized abutments-on the volumetric and linear changes in peri-implant soft tissues, especially when implants are placed subcrestally in healed ridges. This study aims to address that gap through a randomized controlled clinical trial using modern digital tools for volumetric analysis.

Study Objectives:

Primary Objective:

To compare the volumetric changes in peri-implant soft tissue among three different healing abutment designs (standard, wide, and customized) placed over subcrestally positioned bone-level implants in healed ridges.

Secondary Objectives:

To assess the linear changes in gingival margin position and mucosal thickness.

To evaluate the influence of healing abutment design on the stability of the emergence profile.

To explore potential correlations between abutment geometry and soft tissue recession or contour collapse.

To analyze patient-reported outcomes related to esthetic satisfaction and perceived tissue healing.

Study Design:

This is a single-center, randomized, controlled, parallel-group clinical trial with three intervention arms. Thirty adult patients will be recruited and randomly allocated into one of the three study groups (n = 25 per group). All patients will receive a single bone-level dental implant in a posterior maxillary or mandibular healed site, placed 2 mm subcrestally following a one abutment-one time protocol with platform switching.

Study Groups:

Group 1 (Control Group):

Standard cylindrical titanium healing abutment (prefabricated, regular diameter).

Group 2 (Wide Abutment Group):

Prefabricated wide healing abutment with increased diameter for broader mucosal support.

Group 3 (Customized Abutment Group):

Customized healing abutment fabricated in composite using preformed emergence profiles to replicate the ideal emergence profile of the final prosthesis.

All healing abutments will be placed at the time of implant surgery and will not be disconnected during the healing process, in accordance with the one abutment-one time philosophy.

Inclusion Criteria:

Adults aged 18 years or older.

Non-smoking or light-smoking patients (<10 cigarettes/day).

Good general and oral health.

Healed posterior edentulous site requiring a single implant.

Presence of ≥2 mm of keratinized mucosa.

Bone volume sufficient for subcrestal implant placement without grafting.

Willingness to participate and follow the study protocol.

Exclusion Criteria:

Active periodontal or peri-implant disease.

Systemic diseases affecting healing (e.g., uncontrolled diabetes).

Use of bisphosphonates or immunosuppressants.

Pregnancy or lactation.

History of radiation therapy in the head and neck.

Parafunctional habits (e.g., severe bruxism).

Intervention Protocol:

Surgical Procedure:

All implants will be placed 2 mm subcrestally using a guided surgical protocol.

After implant placement, patients will receive the assigned healing abutment (standard, wide, or customized) immediately.

The abutment will remain in place throughout healing and prosthetic phases.

Digital Workflow:

Intraoral scans (STL files) will be obtained at:

T0 (baseline, immediately post-surgery),

T1 (3 months),

T2 (6 months),

T3 (12 months).

The STL files will be superimposed using best-fit alignment algorithms for accurate 3D comparisons.

Tissue Measurement and Analysis:

Soft tissue changes will be measured in terms of:

Volumetric displacement (mm³) using specialized 3D software.

Linear changes in soft tissue thickness and mucosal margin level (mm).

Qualitative heat maps and color-coded deviations will be used to visualize soft tissue gain/loss.

Primary Outcome Measure:

Change in buccal soft tissue volume (mm³) from baseline to 3 months, based on digital 3D superimposition and volumetric analysis.

Secondary Outcome Measures:

Linear change in mucosal thickness (mm) at 3, 6, and 12 months.

Gingival margin displacement (mm) at buccal and interproximal points.

Stability of the emergence profile during provisional and final restoration stages.

Patient-reported esthetic satisfaction using a visual analog scale (VAS).

Statistical Analysis:

Descriptive and inferential statistics will be used. Continuous variables will be analyzed with repeated measures ANOVA or mixed models. Categorical variables will be evaluated using chi-square or Fisher's exact tests. A p-value < 0.05 will be considered statistically significant.

Sample size was calculated to detect a clinically significant difference of 1 mm³ in soft tissue volume change, with a standard deviation of 0.8, α = 0.05, and 80% power, resulting in 10 subjects per group.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. Ethical approval has been or will be obtained from the institutional review board. Informed consent will be obtained from all participants prior to any study-related procedure.

Expected Outcomes and Significance:

This clinical trial aims to clarify how the design of healing abutments-particularly customized CAD/CAM components-affects the healing and dimensional stability of peri-implant soft tissues. Results from this study could support evidence-based decision-making regarding abutment selection in clinical practice, especially in aesthetic-sensitive or high-demand cases. Improved tissue preservation could lead to better prosthetic outcomes and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients requiring a single dental implant in a healed posterior site (maxilla or mandible).
* Presence of at least 2 mm of keratinized mucosa at the implant site.
* Healed alveolar ridge with sufficient bone volume for implant placement without need for guided bone regeneration.
* Good general and oral health, with controlled plaque and bleeding indices.
* Insertion torque ≥ 30 Ncm at the time of implant placement.
* Willingness to comply with study protocol and attend scheduled follow-up visits.
* Signed informed consent.

Exclusion Criteria:

* Smoking more than 10 cigarettes per day.
* Uncontrolled systemic diseases (e.g., uncontrolled diabetes, immunosuppression).
* History of head or neck radiation therapy.
* Current or recent use of bisphosphonates.
* Active periodontal disease or peri-implant infection.
* Severe parafunctional habits (e.g., bruxism, clenching).
* Pregnant or breastfeeding women.
* Previous implant failure at the intended site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Dimensional changes in the peri-implamt soft tissue | Preoperative, the day of the intervention and a follow up until 12 months
  Soft tissue changes will be assessed using digital intraoral scans obtained at baseline, immediately after surgery, and at 3, 6, and 12 months. STL files will be superimposed using 3D analysis software based on stable anatomical landmarks. Volumetric and linear changes will be calculated within defined buccal and interproximal regions of interest (ROIs). Parameters include soft tissue volume (mm³), thickness (mm), and gingival margin displacement. Color-coded deviation maps will visualize contour stability. All measurements will be performed in duplicate by calibrated, blinded evaluators. This method offers accurate, reproducible, and non-invasive assessment of peri-implant soft tissue dynamics.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de València, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez A, Caiazzo A, Valente NA, Toti P, Alfonsi F, Barone A. Standard vs customized healing abutments with simultaneous bone grafting for tissue changes around immediate implants. 1-year outcomes from a randomized clinical trial. Clin Implant Dent Relat Res. 2020 Feb;22(1):42-53. doi: 10.1111/cid.12871. Epub 2019 Dec 3. PMID 31797548
- [Background] Chokaree P, Poovarodom P, Chaijareenont P, Rungsiyakull P. Effect of Customized and Prefabricated Healing Abutments on Peri-Implant Soft Tissue and Bone in Immediate Implant Sites: A Randomized Controlled Trial. J Clin Med. 2024 Feb 2;13(3):886. doi: 10.3390/jcm13030886. PMID 38337580
- [Background] Puisys A, Auzbikaviciute V, Vindasiute-Narbute E, Pranskunas M, Razukevicus D, Linkevicius T. Immediate implant placement vs. early implant treatment in the esthetic area. A 1-year randomized clinical trial. Clin Oral Implants Res. 2022 Jun;33(6):634-655. doi: 10.1111/clr.13924. Epub 2022 Apr 7. PMID 35318752
- [Background] Akin R, Chapple AG. Clinical Advantages of Immediate Posterior Implants With Custom Healing Abutments: Up to 8-Year Follow-Up of 115 Cases. J Oral Maxillofac Surg. 2022 Dec;80(12):1952-1965. doi: 10.1016/j.joms.2022.08.014. Epub 2022 Aug 30. PMID 36155739